CLINICAL TRIAL: NCT04748354
Title: Reshaping the Path Post Hip Fracture in Mild Cognitive Impairment
Brief Title: Reducing Fall Risk Post Hip Fracture in Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Amgen (Industry)
Responsible Party: Principal Investigator, Teresa Liu-Ambrose, Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H19-03812
Record Dates: First submitted 2021-02-01; First posted 2021-02-10 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Hip Fractures; Mild Cognitive Impairment
Keywords: Mobility; Exercise; Fall Risk
MeSH Terms: conditions — Hip Fractures; Cognitive Dysfunction; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Usual care vs. Usual Care with Exercise
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessor and study investigators are blinded to group allocation of participants. Participant cannot be blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Clinical care provided by geriatricians. Each participant will see the geriatrician at baseline and 6 months.
  Interventions: Other: Usual Care
- Usual Care with Exercise (Experimental): Clinical care provided by geriatricians. Each participant will see the geriatrician at baseline and 6 months. In addition, they will receive the Otago Exercise Program, an individualized and home-based program of progressive strength and balance training exercises delivered by a physical therapist.
  Interventions: Behavioral: Otago Exercise Program; Other: Usual Care

INTERVENTIONS:
Behavioral: Otago Exercise Program — An individualized and home-based program of progressive strength and balance training exercises delivered by a physical therapist
  Other Names: Exercise
  Arms: Usual Care with Exercise
Other: Usual Care — Clinical care provided by a geriatrician.

SUMMARY:
Hip fracture is recognized as one of the most serious consequences of osteoporosis, less than half regain pre-fracture independence. 95% of all hip fractures in older adults are due to falls. Thus, reducing fall risk while restoring function post-hip fracture is critical. Many with fall-related hip fractures have cognitive impairment; cognitive impairment increases the risk of falls. The purpose of this 6-month proof-of-concept randomized controlled trial (RCT) is to assess the efficacy of the home-based Otago Exercise Program (OEP) compared with usual care in reducing fall risk among older adults with mild cognitive impairment (MCI) and a fall-related hip fracture.

DETAILED DESCRIPTION:
Hip fracture is recognized as one of the most serious consequences of osteoporosis, less than half regain pre-fracture independence. 95% of all hip fractures in older adults are due to falls. Thus, reducing fall risk while restoring function post-hip fracture is critical. Many with fall-related hip fractures have cognitive impairment and they are less likely to regain pre-fracture level of function than those without cognitive impairment. Cognitive impairment also increase falls risk. It is currently unknown whether exercise is efficacious in reducing fall risk and promoting function among older adults with mild cognitive impairment (MCI) and a fall-related hip fracture. The purpose of this 6-month proof-of-concept RCT is to assess the efficacy of the home-based Otago Exercise Program (OEP) compared with usual care in reducing fall risk among community-dwelling older adults with MCI and a fall-related hip fracture.

ELIGIBILITY:
Inclusion Criteria: 1) aged 65 or older; 2) sustained a fall-related hip fracture in the last 12 months and have returned home; 3) have preserved general cognition as indicated by a Mini-Mental State Examination (MMSE) score = or > 20/30; 4) have subjective memory complaints, determined by interview;22 5) score < 26/30 on the Montreal Cognitive Assessment (MoCA); 6) have an absence of significant functional impairment and no dementia as determined by a physician; 7) are not expected to start, or are stable (i.e., > 3 months) on a fixed dose of anti-dementia medications (e.g., donepezil, galantamine) during the RCT; 8) are expected to live > 12 months (based on the geriatricians' expert opinion); 9) can read, write, and speak English with acceptable visual and auditory acuity; 10) are able to walk 3 meters with or without an assistive device; and 1) provide written informed consent.

Exclusion Criteria: 1) diagnosed with or suspected to have (by the geriatrician) a neurodegenerative disease (e.g., Parkinson's disease) or dementia; 2) had a clinical stroke; or 3) have a history indicative of carotid sinus sensitivity (i.e., syncopal falls).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-05-09 (Actual)

PRIMARY OUTCOMES:
Change in Physiological Profile Assessment | Baseline to 6 Months
  A measure of fall risk (z-score).

SECONDARY OUTCOMES:
Change in Short Physical Performance Battery | Baseline to 3 Months and 6 Months
  A measure of balance and mobility (out of 12 points).
Change in Usual Gait Speed | Baseline to 3 Months and 6 Months
  Gait speed over 4 meters (m/s).
Change in Life Space Assessment | Baseline to 3 Months and 6 Months
  Mobility within a life-space level.
Change in NIH Cognitive Toolbox | Baseline to 3 Months and 6 Months
  Cognitive performance of executive functions.
Change in Digit Symbol Substitute Test | Baseline to 3 Months and 6 Months
  Cognitive performance of processing speed.
Change in Center for Epidemiological Studies Depression Scale | Baseline to 3 Months and 6 Months
  Mood
Change in Positive and Negative Affect Scale | Baseline to 3 Months and 6 Months
  Mood
Change in EQ-5D-5L | Baseline to 3 Months and 6 Months
  Quality of Life
Change in ICE-CAP | Baseline to 3 Months and 6 Months
  Wellbeing
Change in Physical Activity for the Elderly | Monthly from Baseline to 6 Months
  Physical activity over the last 7 days
Total Number of Prospective Falls | Monthly from Baseline to 6 Months
  Self-report of falls using calendars
Change in Activities Specific Balance Confidence | Baseline to 3 Months and 6 Months
  Fall-related self efficacy
Change in Physiological Profile Assessment | Baseline to 3 Months
  A measure of fall risk (z-score); higher z scores indicate higher risk of falls.
Change in Timed Up and Go Test | Baseline to 3 Months and 6 Months
  A measure of functional mobility; greater time for completion indicate poorer performance.
Change in Fried Frailty | Baseline to 3 Months and 6 Months
  A measure of physical frailty
Change in Clinical Frailty Scale | Baseline to 3 Months and 6 Months
  A measure of frailty; higher value indicate more frailty
Change in Pittsburgh Sleep Quality Index | Baseline to 3 Month and 6 Months
  A measure of subjective sleep quality
Change in Rey Auditory Verbal Learning | Baseline to 3 Month and 6 Months
  A measure of episodic memory; higher scores indicate bettter episodic performance.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Liu-Ambrose, PhD, Principal Investigator — University of British Columbia; Larry Dian, MD, Principal Investigator — University of British Columbia; Jennifer C Davis, PhD, Principal Investigator — University of British Columbia; Deborha Jehu, PhD, Principal Investigator — University of British Columbia; Pierre Guy, MD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Vancouver, British Columbia, Canada